CLINICAL TRIAL: NCT00256321
Title: A Phase II Study of Celecoxib/Oxaliplatin/Capecitabine Combination Chemotherapy for Unresectable,Recurrent, or Metastatic Gastric/Gastroesophageal Junction Carcinoma
Brief Title: Celecoxib/Oxaliplatin/Capecitabine for Gastric/Gastroesophageal Junction Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to poor accrual
Sponsor: University of California, Irvine (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Principal Investigator, Chao Family Comprehensive Cancer Center, Cancer Center, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 03-34; 2003-3414 (Other: University of California, Irvine)
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Gastric Carcinoma; Gastroesophageal Junction Carcinoma
Keywords: Gastric Carcinoma; Gastroesophageal junction Carcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Celecoxib/Oxaliplatin/Capecitabine (Experimental): Oxaliplatin 70mg/m2 IV on Days 1 and 8. Capecitabine 1000mg/m2 PO BID from Days 1 through 14. Celecoxib 400mg PO BID from Days 1 through 21.
  1 Cycle = 21 days.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Celecoxib

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 70mg/m2 IV on Days 1 and 8
  Other Names: Eloxatin
Drug: Capecitabine — Capecitabine 1000mg/m2 PO BID from Days 1 through 14.
  Other Names: Xeloda
Drug: Celecoxib — Celecoxib 400mg PO BID from Days 1 through 21.
  Other Names: Celebrex

SUMMARY:
Gastric cancer is the second most common neoplasm in the world. Early diagnosis and surgical resection improve the survival and the chance of cure. Unfortunately, majority of cases are diagnosed at advanced stage, with only 20% of the patients presenting with localized disease. The five-year survival for gastric cancer of all stages remains at a dismal 8%. Chemotherapy has been used for advanced gastric cancer but with unsatisfactory results. Therefore, new approaches are needed for these patients. Among the newer chemotherapy regimens for advanced gastric cancer include a combination of oral 5-Fluoro-Uracil (FU)-based compound called Capecitabine(Xeloda) and Oxaliplatin. A few phase II studies suggest that the combination regimen is active with overall response rates ranging 30-40%. Several preclinical and clinical studies have shown that the expression of cyclooxygenase enzyme II(COX-2) is upregulated in many pre-neoplastic and neoplastic lesions. Furthermore, there appears to be an association with the overexpression of Cox-2 and the invasiveness of cancer and prognosis. Finally, preclinical and clinical studies suggest selective Cox-2 inhibitors can induce apoptosis in gastric cancer cells and retard tumor progression. Therefore, there is a strong rationale for the combination of a selective Cox-2 inhibitor, Celecoxib, with Capecitabine and Oxaliplatin in a therapeutic phase II trial for patients with advanced or recurrent gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically proven, pathologically verified and surgically incurable(unresectable, recurrent, or metastatic) gastric/gastroesophageal junction carcinoma. Gastric lymphoma and Gastrointestinal stromal tumor(GIST) are ineligible for this study. At least 6 unstained paraffin-embedded pathologic specimen slides will be required for the COX-2 expression assays.
* Patient must have bidimensionally measurable disease as defined below. Measurable lesions must be assessed (by physical examination, CT scan, radionuclide scan or plain X-ray) within 30 days prior to registration. The patient's disease status must be completely assessed and reported.

(Measurable Disease: Bidimensionally measurable lesions with clearly defined margins by: 1) Ruler measurement or medical photograph (skin or oral lesion), or plain x ray with at least one diameter .5 cm or greater (bone lesions are not included) or, 2) CT, MRI or other imaging scan with both diameters greater than the distance between cuts of the imaging study, or 3) palpation with both diameters 2 cm or greater.)

* All patients must undergo a CT of abdomen and chest within 30 days prior to registration.
* Patients may have received prior radiation therapy. Radiation therapy must have been completed at least 30 days before registration.
* Patients may have received prior surgery. Prior surgery must have been completed at least 30 days before registration.
* Performance status must be 0-2 according to Southwest Oncology Group Criteria

Exclusion criteria:

* Patients with brain metastases are NOT eligible for this study. It is not mandatory to obtain brain CT or MRI on all patients. However, patients who exhibit neurological symptoms or have pulmonary metastases on radiographic studies must obtain brain CT w/ IV contrast or MRI prior to registration to ascertain the presence of brain metastasis.
* Patients must NOT have received capecitabine or oxaliplatin. Prior use of cisplatin, carboplatin, 5-FU are permitted. Prior systemic therapy must have been completed at least 30 days before registration.
* Pregnant or nursing women are not eligible to participate in this trial because the safe use of these drugs in pregnancy have not been established. Urine pregnancy test must be done prior to the study.
* Patient must NOT have known allergic reaction to sulfonamides
* Patient must NOT have known allergic or other adverse reaction to celecoxib
* Patient must NOT have persistent peripheral neuropathy
* Patient must NOT have known hypersensitivity reactions to 5-FU or platinum
* Patient must NOT have active gastric/duodenal bleeding
* Patient must NOT have had a sensitivity reaction to aspirin or other NSAIDS nonsteroidal antiinflammatory drugs (NSAIDS) [experiencing asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs]

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Response rate of patients with gastric/gastroesophageal carcinoma when treated with celecoxib, oxaliplatin, and capcetabine combination therapy | 18 weeks
  Complete Response (CR) Complete disappearance of all measurable and evaluable disease. No new lesions. No disease related symptoms. No evidence of non evaluable disease, including normalization of markers and other abnormal lab values. All measurable, evaluable and non evaluable lesions and sites must be assessed using the same techniques as baseline.
  Partial Response (PR): Applies only to patients with at least one measurable lesion. Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions. All measurable and evaluable lesions and sites must be assessed using the same techniques as baseline.
  A response rate (RR) is defined as a complete or partial response. RR=CR+PR
Determine time to progression | 18 weeks
  Progression: 50% increase or an increase of 10 CM2 (whichever is smaller) in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, or clear worsening of any evaluable disease, or reappearance of any lesion which had disappeared, or appearance of any new lesion/site, or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer). For "scan only" bone disease, increased uptake does not constitute clear worsening. Worsening of existing non evaluable disease does not constitute progression.

SECONDARY OUTCOMES:
Incidence of treatment-related study adverse events and toxicity according to NCI Common Toxicity Criteria v2.X | 18 weeks
  Toxicity and adverse events are graded on CTC (NCI Common Toxicity Criteria) version 2.X.
Evaluate the expression of the Cox-2 on paraffin-embedded tumor sections from patients enrolled on the study and correlate expression with clinical response | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Randall Holcombe, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States